CLINICAL TRIAL: NCT06067893
Title: Dexmedetomidine as a Pain Management Adjunct in the Pediatric Population Undergoing Posterior Spinal Fusion
Brief Title: Low Dose Dexmedetomidine as a Postoperative Pain Adjunct
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Nichole Doyle (Other)
Responsible Party: Sponsor-Investigator, Nichole Doyle, Physican, M.D., Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00002630
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Spinal Fusion; Adolescent Idiopathic Scoliosis
Keywords: Pain management; Narcotic sparing; Pediatric; Dexmedetomidine
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Patient receives low dose dexmedetomidine infusion in addition to normal post-operative pain management protocol
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): Patient receives normal saline infusion in addition to normal post-operative pain management protocol
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patient receives dexmedetomidine for 48 hours post-operatively
  Arms: Dexmedetomidine
Drug: Normal Saline — Patient receives normal saline for 48 hours post-operatively
  Arms: Control

SUMMARY:
This randomized controlled trial examines whether the addition of a low-dose dexmedetomidine infusion to our current multimodal pain management plan decreases narcotic consumption and reduces side effects in adolescent patients undergoing posterior spinal fusion for idiopathic scoliosis.

DETAILED DESCRIPTION:
Patients will assigned to one of two groups. Either the intervention group where they will receive a dexmedetomidine infusion at 0.2mcg/kg/hr for 24 hours post-operatively or the control group where they will receive a normal saline infusion for 24 hours post-operatively in addition to our hospitals standard pain management protocol. Pain scores will be recorded and patients will fill out a brief questionnaire on POD 1 about their pain control and side effects (pruritus, nausea, vomiting, drowsiness).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic scoliosis
* Undergoing a posterior spinal fusion of at least 5 levels with both thoracic and lumbar involvement

Exclusion Criteria:

* Known allergy to dexmedetomidine or any of the standard medications used intra or post operatively
* Patients with a history of chronic pain currently taking opioids, TCA's, Gabapentinoids
* Medical contraindications to administration of dexmedetomidine, unstable cardiac status, (prolonged Qtc, life threatening arrhythmias, use of digoxin)
* Moya Moya disease

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
narcotic consumption | 48 hours post-operatively
  measuring narcotic consumption in mg/kg per 24 hours in morphine equivalents

SECONDARY OUTCOMES:
Incidence of side effects (nausea, vomiting, pruritus) | 48 hours post-operatively
  Assessing the incidence of side effects (nausea, vomiting, pruritus) using a questionnaire and documented episodes of emesis
Patient safety | 24 hours post-operatively
  Need to discontinue infusion due to over sedation (Ramsey score of 4 or greater), bradycardia (HR <50 sustained on 2 assessments or symptomatic), hypotension (SBP<85 on 2 consecutive assessments or symptomatic). If these HR and SBP safety parameters are not appropriate for a participant based on baseline measurements or medical history new limits will be entered in a nurse communication.

CONTACTS AND LOCATIONS:
Overall Officials: Nichole M Doyle, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified patient data available on request

REFERENCES:
- [Background] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Background] Kaye AD, Chernobylsky DJ, Thakur P, Siddaiah H, Kaye RJ, Eng LK, Harbell MW, Lajaunie J, Cornett EM. Dexmedetomidine in Enhanced Recovery After Surgery (ERAS) Protocols for Postoperative Pain. Curr Pain Headache Rep. 2020 Apr 2;24(5):21. doi: 10.1007/s11916-020-00853-z. PMID 32240402
- [Background] Naduvanahalli Vivekanandaswamy A, Prasad Shetty A, Mugesh Kanna R, Shanmuganathan R. An analysis of the safety and efficacy of dexmedetomidine in posterior spinal fusion surgery for adolescent idiopathic scoliosis: a prospective randomized study. Eur Spine J. 2021 Mar;30(3):698-705. doi: 10.1007/s00586-020-06539-9. Epub 2020 Jul 21. PMID 32696258
- [Background] Panchgar V, Shetti AN, Sunitha HB, Dhulkhed VK, Nadkarni AV. The Effectiveness of Intravenous Dexmedetomidine on Perioperative Hemodynamics, Analgesic Requirement, and Side Effects Profile in Patients Undergoing Laparoscopic Surgery Under General Anesthesia. Anesth Essays Res. 2017 Jan-Mar;11(1):72-77. doi: 10.4103/0259-1162.200232. PMID 28298760